CLINICAL TRIAL: NCT03885310
Title: Gastrointestinal Drug-Coated Balloon for the Treatment of Symptomatic Recurrent Benign Esophageal Stricture
Brief Title: INGEST I Pilot Study
Acronym: INGEST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GIE Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR2001
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Esophageal Stricture
MeSH Terms: conditions — Esophageal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DCB Treatment (Experimental): Stricture patients treated by DCB
  Interventions: Device: GIE Drug Coated Balloon

INTERVENTIONS:
Device: GIE Drug Coated Balloon — The GIE DCB is a balloon catheter with a 3 stage inflatable balloon coated with a proprietary coating containing the drug and carriers.

SUMMARY:
INGEST I Pilot study is a feasibility study for evaluating the safety and efficacy of DCBs.

DETAILED DESCRIPTION:
The study is designed to determine the safety and effectiveness of drug coated balloon (DCB) treatments on esophageal stricture.

Up to 30 subjects are planned to be enrolled and treated with the study device at up to 5 clinical sites outside of US. Subjects will be followed up post-treatment to one year and then annually for up to 5 years. The annual follow up after the first year is optional.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 80 years.
2. Benign esophageal stricture with diameter less than 10 mm (barium esophagram).
3. Dysphagia score of 2 to 4 (Ogilvie Dysphagia Score).
4. Recurrent stricture after at least 2 previous balloon/bougie dilation or stricturotomy sessions.
5. Stricture total length ≤ 7 cm. Tandem or adjacent strictures are allowed if the strictures are caused by the same underlining disease.
6. Ability to undergo periodic endoscopic follow-up.
7. Voluntary participation and provided written informed consent.

Exclusion Criteria:

1. Pregnancy or breastfeeding or plan to get pregnant in next 12 months.
2. Contraindication to endoscopy, anesthesia or deep sedation.
3. Benign esophageal stricture due to extrinsic esophageal compression.
4. Currently required chest radiation therapy.
5. Malignant esophageal stricture.
6. Stricture total length > 7 cm or esophageal strictures at multiple locations where the total stricture length exceeds 7 cm
7. Dysphagia related to primary motility disorders, such as achalasia, diffused esophageal spasm, ineffective esophageal motility (IEM), hypertensive lower esophageal sphincter, etc.
8. Active erosive esophagitis.
9. Present esophageal ulceration, perforation, leak, fistula, or varices.
10. Concurrent gastric and/or duodenal obstruction.
11. Active systemic infection.
12. Allergy to paclitaxel or any components of the delivery system.
13. Severe coagulation disorders or current use of anticoagulant for comorbidities.
14. Chronic steroid use for any medical conditions unless subject is willing to undergo a 4-week washout and discontinue steroid use.
15. Received steroid injections into target stricture in the last 4 weeks
16. Intolerant to proton pump inhibitors.
17. Life expectancy of less than 12 months.
18. Unwilling or unable to comply with the follow-up study requirements.
19. Lacking capacity to provide informed consent.
20. Concurrent medical condition that would affect the investigator's ability to evaluate the patient's condition or could compromise patient safety, such as recent myocardial infarction, severe pulmonary disease, bleeding diathesis, large thoracic aneurysm, recent laparotomy, pharyngeal or cervical deformity, etc.
21. Currently participation in another pre-market drug or medical device clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-02-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incident of serious balloon dilation-related complications | 30 days
  Adverse events such as perforation, bleeding requiring intervention, severe pain during swallowing, infection requiring hospitalization or IV antibiotics, dysphagia requiring re-intervention at determined by the attending physician

SECONDARY OUTCOMES:
Numbers of additional esophageal dilation procedures | 30 days, 3 months, 6 months, and 12 months
  Repeat stricture treatments
Time to first dysphagia symptom recurrence | 30 days, 3 months, 6 months, and 12 months
  Ogilvie Dysphagia Score will be used to assess subject's dysphagia symptom changes at follow-ups. The date of the first reported occurrence of dysphagia symptom will be used to derive the time to first dysphagia symptom recurrence.
Improvement in dysphagia score | 30 days, 3 months, 6 months, and 12 months
  Ogilvie Dysphagia Score will be used to assess subject's dysphagia symptom changes at follow-ups. The scores at each follow-up will be compared to the score at baseline.
Esophageal stricture diameter | 30 days, 3 months, 6 months, and 12 months
  Endoscopy and esophagography will be conducted to measure the internal caliber of the esophagus. Results will be reported in millimeters.
Technical success | Time of procedure
  Successful delivery of the drug coated balloon to the target stricture, balloon inflation to the desired pressure, balloon deflation and withdraw without device malfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Wang, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Adventista Hospital, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang KK, Schorn I, Adorno C. Development and initial clinical experience with a paclitaxel-coated balloon for the treatment of benign difficult esophageal strictures. IGIE. 2023 Sep 17;2(4):399-407. doi: 10.1016/j.igie.2023.09.004. eCollection 2023 Dec. PMID 41646070